CLINICAL TRIAL: NCT06508918
Title: The Effect of Central Sensitization on the Treatment Success of Ultrasound-Guided Caudal Epidural Steroid Injection in Radicular Pain in Patients With Failed Back Surgery Syndrome
Brief Title: The Effect of Central Sensitization in Radicular Pain in Patients With Failed Low Back Surgery Syndrome
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 03.03.2023.375
Record Dates: First submitted 2023-04-09; First posted 2024-07-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Herniated Disc; Failed Back Surgery Syndrome
MeSH Terms: conditions — Intervertebral Disc Displacement; Failed Back Surgery Syndrome | interventions — Betamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1 (with central sensitization): Group: group 1 (with central sensitization) 8 mg betamethasone, 3 cc bupivacaine, 5 cc serum will be injected in the neck, and caudal force pressure, pressure pain thresholds will be evaluated with a manual algometer, accompanied by ultrasonography.
  Group: group 2 (without central sensitization) 8 mg betamethasone, 3 cc bupivacaine, 5 cc serum will be injected in the neck, and caudal force pressure, pressure pain thresholds will be evaluated with a manual algometer, accompanied by ultrasonography.
  Interventions: Drug: Betametasona
- group 2 (without central sensitization): Group: group 1 (with central sensitization) 8 mg betamethasone, 3 cc bupivacaine, 5 cc serum will be injected in the neck, and caudal force pressure, pressure pain thresholds will be evaluated with a manual algometer, accompanied by ultrasonography.
  Group: group 2 (without central sensitization) 8 mg betamethasone, 3 cc bupivacaine, 5 cc serum will be injected in the neck, and caudal force pressure, pressure pain thresholds will be evaluated with a manual algometer, accompanied by ultrasonography.
  Interventions: Drug: Betametasona

INTERVENTIONS:
Drug: Betametasona — pressure pain threshold values of the most painful area will be recorded with a manual algometer
  Other Names: baseline brand algometer

SUMMARY:
The Effect of Central Sensitization in Radicular Pain in Patients with Failed Low Back Surgery Syndrome on Treatment Success of Ultrasound-Guided Caudal Epidural Steroid Injection

DETAILED DESCRIPTION:
Low back pain is a very common clinical picture that has a tremendous social, financial and psychological impact on the patient's life. It is a worldwide problem with a global incidence of 9.4% and causes more disability than any other condition in the world. The percentage of adults who experience chronic low back pain throughout their lives ranges from 51% to 84% . As the population ages, the incidence of surgery for low back pain increases dramatically; the number of lumbar fusions increased by 170% from 1998 to 2008. Failed back surgery syndrome (FBSS) has been reported to affect 10 to 40% of patients following spine surgery, but estimating the incidence of FBSS is difficult due to the wide scope of its definition and heterogeneous etiology. Failed back surgery syndrome (FBSS) is defined by the International Association for the Study of Pain as "lumbar spinal pain of unknown origin that persists despite surgical intervention or occurs after surgical intervention for pain in the same topographic region". Pain may occur after surgery, surgery may exacerbate existing pain or not adequately improve it. Patients with FBSS have undergone one or more surgical interventions that do not cure long-standing chronic low back pain and pain, with or without radicular symptoms. Its etiology is complex and it is a condition with many factors that predispose patients to chronic pain. Epidural fibrosis, perineural scars, acquired stenosis, recurrent disc herniation or pain of the sacroiliac/facet joints are thought to play a role in the etiology of FBSS. Pain in the leg likely indicates nerve compression from stenosis, epidural fibrosis, or disc herniation, while low back pain is more common in facet joint arthropathy, sacroiliac joint problems, or myofascial etiologies. For the failed back surgery syndrome patient, physical examination is usually not helpful in identifying a specific aetiology of pain, but may reveal several suggestive findings. Symptoms from spinal stenosis are usually exacerbated by spinal extension and relieved by flexion. On the other hand, pain from disc herniation causes a positive straight leg raise test. Loss of strength or sensation in the lower extremities can help to understand which nerve roots are affected. Other tests may be used to elucidate the etiology of failed back surgery syndrome and differentiate it from other causes of low back pain. Erythrocyte sedimentation rate and C-reactive protein can be used to evaluate possible infection, especially in patients with structural symptoms or susceptibility to infection. Diagnostic nerve blocks can diagnose specific etiologies of FBSS, such as facet joint arthropathy (medial bundle blocks), sacroiliac joint pain (lateral bundle branch blocks and intra-articular injection), and foraminal stenosis (transforaminal epidural and selective unilevel blocks) and roots associated with the patient's symptoms. can define. MRI with and without gadolinium contrast remains the gold standard imaging modality for failed back surgery syndrome, as it can perfectly detect soft tissue abnormalities such as epidural fibrosis and disc herniation. Contrast is particularly indicated in patients with a history of disc herniation surgery. A panel of international spine surgeons, neurosurgeons, and pain specialists with a special interest in FBSS established the Chronic Low Back and Leg Pain (CBLP) network to address the challenges and barriers in the clinical management of FBSS patients, creating a collaborative interdisciplinary body. The definition of FBSS proposed by the CBLP network is based on the assumption that no further spine surgery is required after an appropriate somatic, radiological, and psychosocial assessment. The key elements for the definition of FBSS can be summarized in 4 aspects:

1. There is low back and/or leg pain that persists for at least 6 months after the last spine surgery
2. Patient has undergone a comprehensive clinical and radiological evaluation
3. There is no clear surgical target consistent with the symptoms revealed on clinical examination and imaging
4. There is an interdisciplinary consensus that additional surgical intervention (decompression and/or fusion) is not appropriate.

Despite its adverse effects on patients and its relative prevalence in the spine surgery population, few high-quality randomized studies have investigated the treatment of FBSS. Treatments for FBSS are generally divided into conservative (physical therapy or drug therapy) and aggressive (interventional or surgical) management. Conservative treatment should always be the first choice before invasive techniques in patients without an indication for emergency surgery. Various studies have shown that caudal epidural steroid injection (CESI) is an effective method in patients with FBSS who do not respond to conservative pain relief treatments . Çelenlioğlu A. et al. investigators compared the success of transforaminal epidural steroid injection (TFESI ) and CESI treatment in patients who developed FBSS after single-level discectomy. In two prospective randomized studies, both CESI and TFESI (transforaminal epidural steroid injection) were found to be effective and safe in treatment. CESI has been shown to be the safest and simplest ESI with a low complication rate, including dural puncture and other side effects, compared to other injection methods. Yoon et al. reported a success rate of 94% with US-guided caudal blockade. In a study conducted by Akkaya et al. when ultrasound and fluoroscopy-guided caudal epidural steroid injection (CESI) were compared to patients with FBSS, a decrease in both pain and ODI (oswestry disabilite index)scores was achieved in both groups at 3-month follow-up, and CESI was found to be effective in the treatment of FBSS. has been reported. In a prospective randomized controlled study comparing the treatment success of caudal epidural steroid injection with ultrasonography (USG) and fluoroscopy in postlaminectomy patients, no difference was found between the two groups in terms of complications, while the patients in the fluoroscopy group felt more pain during the procedure than the patients in the USG group. Despite correct needle localization and drug injection under fluoroscopy guidance, radiation is still a serious risk for both patient and responder. The use of USG in caudal epidural injections protects from radiation exposure, and is a safe and rapid method for locating the sacral hiatus and guiding the needle. Color Doppler USG can view intravenous injections. Tsui et al. reported that the color Doppler feature of USG could confirm whether the injected drug was diffused to the caudal area. Injection of fluid into the epidural space causes turbulent flow, which appears as a burst of color, while intrathecal injection indicates the absence of color flow Doppler signal. Although the precise pathophysiological process of FBSS remains unclear, growing evidence suggests that widespread pain distribution, hyperalgesia, and disproportionate pain intensity symptoms, which are also common in other chronic pain-related diseases (e.g., fibromyalgia, tension-type headache, and nonspecific chronic low back pain), are a potential risk factor. predicts that central sensitization may develop. The International Association for the Study of Pain (IASP) defined CS in 2011 as "the increased response of nociceptive neurons in the central nervous system to normal or sub-threshold afferent inputs." Anxiety about pain, restriction of daily activities, quality of life and the stress associated with it lead to depression over time and thus a vicious cycle of "pain-anxiety-depression" begins. Altered central pain modulation may be involved in the pathogenesis of FBSS. Unfortunately, only a few studies have investigated the presence of central sensitization, although it may guide the treatment of patients with FBSS. Central amplification of pain may contribute to both chronic low back pain intensity and disability in FBSS patients. Therefore, targeted therapies should consider functional changes in the central nervous system of FBSS patients, and treatment modalities that can weaken central sensitization (eg, cognitive-targeted exercise therapy, pharmacotherapy, spinal cord stimulation) may be beneficial in the treatment of FBSS. Our aim is to reveal the relationship between FBSS and central sensitization proportionally, keeping in mind that central sensitization may develop in post-spinal surgery patients with ongoing pain, to prevent the formation of a vicious circle of chronic pain with its early detection and treatment, and to prevent the formation of a vicious circle of chronic pain. Moreover, caudal epidural steroid injection with USG does not have radiation exposure and it is advantageous and beneficial. Since it is a reliable method, investigators aim to determine its effectiveness in patients with FBSS. As far as investigators know, such a study has not been reported before in the literature, investigators hope that investigators will contribute to the literature.

ELIGIBILITY:
Inclusion criteria:

* 18-75 years old
* Meeting the diagnostic criteria for failed back surgery syndrome
* Radicular pain that begins any time after surgery and lasts for at least 6 months
* Epidural fibrosis and/or disc herniation at the L5 and/or S1 vertebral level on contrast-enhanced MR imaging
* Nrs equal to or greater than 4
* Conservative methods are ineffective
* Volunteer

Exclusion Criteria:

* Acute or chronic uncontrolled medical illness
* Lumbar localization pathologies
* Isolated axial low back pain
* History of lumbar stabilization or non-microdiscectomy lumbar surgery
* History of adverse statements against local anesthesia or steroids being pregnant or breastfeeding
* Stories on the injectables to be administered bleeding diet
* Not wanting to participate in the research

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-75 who have had unsuccessful back surgery and who have had low back and leg pain for at least 6 months that started in the same region before the surgery
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale /NRS | 3rd months
  At least 50 percent improvement in Numeric Rating Scale (NRS more than fifty percent reduction indicates greater improvement. The nrs score is scored from 0 to 100. Higher scores are associated with more pain.)

SECONDARY OUTCOMES:
Improvements in Douleur Neuropathique 4 Questions | 3rd month
  Douleur Neuropathic 4 (DN4) is a scale that evaluates the patient's neuropathic symptoms with 4 questions. On the scale with a total score of 10, those who score above 4 indicate the presence of neuropathic pain.
Improvements in Beck's Depression Inventory | 3rd month
  Beck Depression Inventory the questionnaire consists of a total of 21 questions, each with four options. The total score is calculated by scoring each option in the range of 0-3. In scoring, 0-9 is interpreted as normal, 30-63 as severe depression.
Improvements in Oswestry Disability Index | 3rd month
  The Oswestry Disability Index the maximum score is "100", the minimum score is "0". As the total score increases, the level of disability also increases
Improvements in Central Sensitization inventory | 3rd month
  scored between 0-100 points. The higher the patient's score, the more CS-related symptoms are considered to be.
Improvements in Pressure Pain Thresold values | 3rd month
  The value at which the feeling of pressure turns into a feeling of pain was recorded with a manual algometer. If patients fail to report pain at a pressure of 10 kg/cm2 on pressure pain threshold (PPT) measurements, the test will be stopped and this value will be recorded as PPT.

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Şencan, Principal Investigator — Marmara Universty
Locations (2):
- Turkey (Türkiye) (2):
  - Mamara Üniversitesi Tıp Fakültesi, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul

DOCUMENTS (1):
  • Study Protocol (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT06508918/Prot_000.pdf